CLINICAL TRIAL: NCT06967714
Title: Disentangling the Variability of Exercise-induced Hypoalgesia: the Role of Circulatory Compounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EIH-VAR
Record Dates: First submitted 2025-04-22; First posted 2025-05-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: exercise-induced hypoalgesia; mechanisms; pain; exercise
MeSH Terms: conditions — Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Withi-subject desing. Participants will complete three experimental sessions. In the first session, they will be asked to complete a set of questionnaires and to do a maximal exercise test. The next two sessions will be identical and will consist in blunt pressure sensitivity assessment-before (T0), immediately after (T1), and 45 min after (T2) a 25 min cycling exercise-at body parts involved (lower limb) and non-involved (upper limb, immobilized) in the exercise. Venous blood samples will be collected concomitantly to the sensory testing procedure.
Masking Description: * Participant will be masked to study hypotheses
  * Outcome assessor/Investigator will be masked to sensory tests results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Participants will complete three experimental sessions. In the first session, they will be asked to complete a set of questionnaires and to do a maximal exercise test. The next two sessions will be identical and will consist in blunt pressure sensitivity assessment-before (T0), immediately after (T1), and 45 min after (T2) a 25 min cycling exercise-at body parts involved (lower limb) and non-involved (upper limb, immobilized) in the exercise. Venous blood samples will be collected concomitantly to the sensory testing procedure.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 25 min cycling exercise at 75% of hear rate reserve. Physical use of one upper-limb will be restricted with a sling.

SUMMARY:
Physical exercise is increasingly recognized as an effective treatment for chronic pain. Studies in humans and animals have shown that a single session of exercise induces a reduction of sensitivity to experimental painful stimuli lasting up to 45 minutes. In a recent study conducted in our laboratory, we found (1) that this exercise- induced hypoalgesia (EIH) is mainly driven by local changes in muscle nociceptor sensitivity within exercising muscles and (2) that EIH is consistent at a group level but fluctuates across sessions within participants. The first aim of this project is to uncover the mechanism(s) that drive EIH by investigating whether processes that could contribute to an exercise-induced change in muscle nociceptor sensitivity match the fluctuating pattern of EIH. Specifically, we will assess the possible involvement in EIH of the endocannabinoid system (eCB), Kynurenic acid (KynA, a circulating myokine that transiently increases after exercise), and β -endorphins (βE). Using a sample of 90 healthy males and females aged 18 to 30 years, we will measure sensitivity to blunt pressure stimuli before, immediately after, and 45 min after a 25-min cycling exercise to assess muscle nociceptor sensitivity at exercising (rectus femoris muscle) and non-exercising (ventral forearm) muscles. Blood samples will be collected at these time-points to measure plasma levels of eCBs, βE, and KynA. In addition, the effect of sex on EIH is controversial: some studies report no differences between males and females, while others report a greater effect in males or in females. Therefore, a secondary aim of this study is to explore potential sex differences in the manifestation and underlying mechanism(s) of EIH.

ELIGIBILITY:
Inclusion Criteria:

* Males, or females using hormonal contraception since ≥ 3 months.
* Aged between 18 and 30 years.
* Ability to provide written informed consent.
* Fluency in French or English.
* BMI between 17 and 30 kg/cm2.

Exclusion Criteria:

* Regular tobacco use (> 1/month)
* Not willing or able to abstain from alcohol, recreational drugs, coffee, or tea from 24 hours prior to each experimental session.
* Not willing or able to restrain from physical activity > 24h prior to each experimental session, and to be in a fasted state on the day of each experimental session.
* Any evidence for neurological, cardiovascular, respiratory, inflammatory, endocrine, psychiatric, oncological, rheumatological conditions on direct questioning.
* Presence of any medical devices (e.g., cardiac pacemaker) implants or prothesis unless it is beyond discussion that these will not put the subject's safety during the study at risk and will not interfere with the results of the study.
* Any chronic pain condition or recent history thereof (i.e., within the preceding 2 years).
* Wounds or skin alteration on testing sites.
* Surgery < 12 months.
* Any drug intake in the past 2 weeks including antibiotics, herbal medicines and other remedies except the following drugs that will be allowed up to 48 hours prior to the experiments: oral paracetamol or ibuprofen for a self-limiting condition (e.g. toothache, bruise). Oral antihistaminics and nasal aerosol and topical treatments for seasonal allergy up to 1 week before the experimental session.
* Any physical activity contraindication.
* Pregnancy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pressure pain threshold | At each experimental experimental session (2 in total): before (T0), immediately after (T1), and 45 min (T2) after the intervention (cycling exercise).
  The investigators will use blunt pressure to preferentially activate the mechano-sensitive deep-tissue nociceptors. The stimuli will be delivered with a manual digital algometer with a contact surface area of 1cm2 (FPIX; Wagner Instruments, Greenwich, USA) connected to a laptop computer through a USB-serial port. A bespoke Matlab (The Mathworks, USA, mathworks.com) script will provide visual feedback of the force application rate to the examinator, while blinding him to the final threshold value. The participants will be asked to report the first onset of pain by pressing on a keyboard key, defining the pressure pain threshold (PPT). The procedure is safe, and there are no side effects to the stimulation

SECONDARY OUTCOMES:
Plasmatic levels of endocannabinoids | At each experimental experimental session (2 in total): before (T0), immediately after (T1), and 45 min (T2) after the intervention (cycling exercise).
  Blood samples will be collected after catheterization of an upper limb vein. The investigators will collect blood samples before, immediately after, and 45 min after exercise (at each session) to investigate potential EIH contributors. Specifically,the plasmatic levels of the endocannabionid (anandamide and 2-Arachidonoylglycerol) will be measured.
Plasmatic level of Kynurenic acid | At each experimental experimental session (2 in total): before (T0), immediately after (T1), and 45 min (T2) after the intervention (cycling exercise).
  Blood samples will be collected after catheterization of an upper limb vein. The investigators will collect blood samples before, immediately after, and 45 min after exercise (at each session) to investigate potential EIH contributors. Specifically, plasmatic levels of kynurenic acid will be measured.
Plasmatic level of and beta-endorphin | At each experimental experimental session (2 in total): before (T0), immediately after (T1), and 45 min (T2) after the intervention (cycling exercise).
  Blood samples will be collected after catheterization of an upper limb vein. The investigators will collect blood samples before, immediately after, and 45 min after exercise (at each session) to investigate potential EIH contributors. Specifically, the plasmatic levels of beta-endorphins will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Institute of neuroscience, Brussels, Belgium, Belgium

IPD SHARING:
Plan to Share IPD: No